CLINICAL TRIAL: NCT06629688
Title: The Effect of Parenterally Administred Semaglutide on Intestinal Iron Absorption in Individuals With Type 2 Diabetes Mellitus
Brief Title: Semaglutide and Intestinal Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Petra Meliš, Principal Investigator, University Hospital Dubrava
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sema-iron
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus Type 2; Iron Absorption
Keywords: type 2 diabetes mellitus; semaglutide; iron; oral iron absorption test
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Patients between the ages of 45 and 65 with poorly controlled T2DM (HbA1c ≥ 7%) who were candidates for treatment intensification and beginning of parenterally administered semaglutide were eligible to participate in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T2DM subjects before and at week 10 of semaglutide therapy (Experimental): Patient demographic and clinical data was collected and entered into a database made specifically for the study. The patients were examined, and their vital signs and body measures were recorded. Before the introduction of semaglutide therapy all participants completed an oral absorption iron test (OIAT). As described in previous studies, OIAT was conducted in an outpatient setting. Following the initial OIAT therapy with semaglutide was started. Each subject received parenterally administered one-weekly semaglutide. To enhance glycaemic control, the therapy was up-titrated every four weeks. Initially, the dose was set at 0.25 mg once a week, four weeks later, it was raised to 0.5 mg once weekly, and four weeks after that, it was increased to 1 mg once weekly. After reaching the maximum maintenance dosage of 1 mg for two weeks, each T2DM patient completed a follow-up OIAT at week 10 of the study. Data from the first and subsequent OIATs were analysed statistically.
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Patient demographic and clinical data was collected and entered into a database made specifically for the study. The patients were examined, and their vital signs and body measures were recorded. Before the introduction of semaglutide therapy all participants completed an oral absorption iron test (OIAT). As described in previous studies, OIAT was conducted in an outpatient setting. Following the initial OIAT therapy with semaglutide was started. Each subject received parenterally administered one-weekly semaglutide. To enhance glycaemic control, the therapy was up-titrated every four weeks. Initially, the dose was set at 0.25 mg once a week, four weeks later, it was raised to 0.5 mg once weekly, and four weeks after that, it was increased to 1 mg once weekly. After reaching the maximum maintenance dosage of 1 mg for two weeks, each T2DM patient completed a follow-up OIAT at week 10 of the study. Data from the first and subsequent OIATs were analysed statistically.

SUMMARY:
Semaglutide belongs to a group of long-acting glucagon-like peptide 1 receptor agonists (GLP-1). Disorders in iron absorption have been linked to numerous medication, dietary, and nutrient interactions thus far. The study aimed to determine whether there is an effect of concomitant parenteral administration of semaglutide and oral iron preparations on iron absorption in patients with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) affects over 537 million people worldwide, making it a major chronic and progressive health problem among adults. Novel approaches to managing T2DM have been developed as a result of medical advancements. Glucagon-like peptide-1 receptor agonists (GLP-1 RAs) are appealing options for the treatment of T2DM, since they efficiently reduce body weight and haemoglobin A1C with a minimal risk of hypoglycaemia.

Semaglutide, a long-acting GLP-1 RA, has a very high structural homology with endogenous GLP-1, high binding affinity to albumin, and resistance to degradation by the intestinal enzyme dipeptidyl peptidase-4. Because of these characteristics and his extended half-life, it can be used once weekly. Similar to all other GLP-1 RAs, semaglutide decreases gastrointestinal motility and slows stomach emptying. Delay in stomach emptying and intestinal motility can interfere with vitamin, mineral, and drug absorption. Iron is one of the essential micronutrients in the human body. On average, 10 - 20 mg of iron is consumed daily through food, but only 1 - 2 mg of iron is absorbed in the duodenum and the first section of the small intestine. It has been shown that drugs which decrease gastrointestinal motility can interfere with iron absorption. However, the relationship between parenteral semaglutide administration and intestine iron absorption has not been the subject of any prior studies. Thus, this study aimed to determine whether there is an effect of parenteral administration of semaglutide on iron absorption in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* T2DM patients
* ages between 45 and 65
* with poorly managed T2DM (HbA1c ≥ 7%)
* who are candidates for treatment intensification and beginning of parenterally administered semaglutide

Exclusion Criteria:

* hypersensitivity to GLP-1 RAs,
* adequately controlled with current glucose-lowering medications,
* already treated with GLP-1 RA,
* type 1 diabetes mellitus or any other form of diabetes,
* hemochromatosis,
* iron deficiency anaemia,
* sideropaenia,
* severe chronic illnesses,
* malignant neoplasms of any site,
* chronic infectious diseases,
* chronic rheumatic inflammatory diseases,
* malabsorption syndrome,
* inflammatory bowel disease,
* history of gastrointestinal tract reduction surgery,
* medications that interfere with absorption,
* perimenopausal women

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
General objective | 10 weeks
  Number of T2DM participant that will have reduction in intestinal iron absorption after the semaglutide administration

SECONDARY OUTCOMES:
Specific objectives | 10 weeks
  Correlation between serum ferritin levels prior to the OIAT and the degree of iron absorption during semaglutide administration in patients with T2DM.

OTHER OUTCOMES:
Sex differences | 10 weeks
  Sex-dependent difference in intestinal iron absorption with the administration of semaglutide in patients with T2DM.

CONTACTS AND LOCATIONS:
Overall Officials: Srećko Marušić, MD, PhD, Principal Investigator — UH Dubrava
Locations (1):
- University hospital Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided